CLINICAL TRIAL: NCT07372573
Title: Effectivenes of Pressurized Meter Dose Inhaler (PMDI) Versus Dry Powder Inhaler (DPI) in Delivering Inhaled Corticosteroid and Long Acting Beta Agonist Among Patients With Uncontrolled Asthma in a Tertiary Care Hospital.
Brief Title: Pressurized Meter Dose Inhaler V/S Dry Powder Inhaler
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Laiba Qamar, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #PMDIDPI#
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Asthma (Diagnosis)
Keywords: Asthma; Pressrized Meter Dose inhaler; Dry powder Inhaler; long acting beta Agonist; inhaled corticosteroid
MeSH Terms: conditions — Asthma; Disease | interventions — Dry Powder Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Patients in this arm will receive a fixed-dose combination of inhaled corticosteroid and long-acting beta agonist (budesonide/formoterol) via a pressurized metered dose inhaler. The prescribed dose will be 200/6 µg per puff, two puffs twice daily, delivering a total daily dose of 800/24 µg. This arm evaluates the effectiveness of aerosol-based drug delivery requiring hand-breath coordination.
  Interventions: Device: Pressurized Metered Dose Inhaler (pMDI)
- Group B (Active Comparator): Patients in this arm will receive the same fixed-dose combination of budesonide/formoterol via a dry powder inhaler at a dose of 400/12 µg per puff, one puff twice daily, achieving the same total daily dose of 800/24 µg. This arm assesses the effectiveness of breath-actuated powder-based drug delivery.
  Both arms use equivalent drug molecules and doses, with the inhaler device being the only variable, allowing direct comparison of device-related effectiveness in uncontrolled asthma.
  If you want, I can also write this in tabular form or CPSP RTMC-preferred wording.
  Interventions: Device: Dry Powder Inhaler

INTERVENTIONS:
Device: Pressurized Metered Dose Inhaler (pMDI) — Participants allocated to this group will be treated with a combination of inhaled corticosteroid and long-acting beta agonist in the form of budesonide/formoterol 200/6 micrograms per actuation delivered via a pressurized metered dose inhaler. Patients will be instructed to take two puffs twice daily, resulting in a total daily dose of 800 micrograms of budesonide and 24 micrograms of formoterol. This intervention evaluates medication delivery through an aerosolized spray that requires proper coordination between actuation and inhalation.
  Arms: Group A
Device: Dry Powder Inhaler — articipants in this group will receive the same combination therapy of budesonide/formoterol 400/12 micrograms per inhalation administered through a dry powder inhaler. The prescribed regimen will be one inhalation twice daily, providing an equivalent total daily dose of 800 micrograms of budesonide and 24 micrograms of formoterol. This intervention assesses drug delivery via a breath-activated powder formulation, where adequate inspiratory effort is required for optimal drug deposition.
  Arms: Group B

SUMMARY:
This study compares two commonly used inhalation devices in asthma management. It focuses on evaluating how effectively PMDIs and DPIs deliver the same combination of inhaled corticosteroids and long-acting beta agonists in patients whose asthma remains poorly controlled despite treatment. The study is conducted in a tertiary care hospital setting, emphasizing real-world clinical practice and aiming to determine whether device choice influences asthma control outcomes.

DETAILED DESCRIPTION:
Asthma is a common chronic respiratory disease, and despite advances in therapy, a significant proportion of patients remain poorly controlled. Inhaled corticosteroids (ICS) combined with long-acting beta agonists (LABA) are the cornerstone of asthma management; however, the effectiveness of treatment is highly dependent on the inhalation device used. Pressurized metered dose inhalers (pMDIs) and dry powder inhalers (DPIs) are the most widely used devices, yet their relative effectiveness in real-world clinical practice remains debated, particularly in resource-limited settings.

This randomized controlled trial aims to compare the effectiveness of pMDI versus DPI in delivering equivalent doses of ICS/LABA among patients with uncontrolled asthma attending the Pulmonology Outpatient Department of Services Hospital Lahore. A total of 210 patients aged 14-60 years with uncontrolled asthma, defined by an Asthma Control Questionnaire (ACQ) score ≥3 despite baseline therapy, will be enrolled using non-probability consecutive sampling and randomized into two groups. Both groups will receive an equivalent total daily dose of budesonide/formoterol (800/24 µg), administered either via pMDI or DPI.

Patients will be followed for eight weeks with assessments at baseline, four weeks, and eight weeks. The primary outcome will be improvement in asthma control measured by reduction in ACQ score, while secondary outcomes include frequency of asthma exacerbations. Data will be analyzed using SPSS version 25, with appropriate statistical tests applied to compare outcomes between groups.

The findings of this study are expected to clarify whether inhaler device choice significantly influences asthma control. This will help distinguish true treatment-resistant asthma from poor control due to device-related factors and guide clinicians in selecting the most effective inhalation device for improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

Age 14 to 60 years

Both genders

All patients with symptoms of uncontrolled asthma

Exclusion Criteria:

Patients with coexistent fungal sensitization (confirmed with peripheral eosinophil count and serum IgE)

Patients with coexistent Allergic Bronchopulmonary Aspergillosis (ABPA) (confirmed with HRCT and serum IgE)

Patients with coexistent COPD (confirmed on spirometry)

Patients with Hypersensitivity Pneumonitis

Patients with coexistent Interstitial Lung Disease (ILD) (confirmed on spirometry)

Patients with coexistent cardiac asthma secondary to heart failure (diagnosed on echocardiography)

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Questionnaire (ACQ) score | 8 weeks
  The primary outcome of this study is improvement in asthma control, assessed by the change in Asthma Control Questionnaire (ACQ) score from baseline to 8 weeks after intervention. Effectiveness will be determined by a reduction in ACQ score compared to the baseline value, reflecting better symptom control with the assigned inhaler device.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No